CLINICAL TRIAL: NCT06981026
Title: The Effectiveness of Telemedicine Monitoring Prehabilitation in Prostate Cancer Patients Undergoing Radical Prostatectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Olomouc (Other)
Collaborators: Mobilní fyzioterapie s.r.o. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OP JAK ITI VZ 2; CZ.02.01.01/00/23_021/0008829 (Other Grant/Funding Number: Operational Programme Jan Ámos Komenský financed by the European Union (EU) and the State Budget of Czech Republic)
Record Dates: First submitted 2025-03-18; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Prostatectomy; Prehabilitation; Telemedicine
Keywords: Prostatectomy; Physiotherapy; Telemedicine; eHealth; Oncology; Prehabilitation; Rehabilitation
MeSH Terms: conditions — Neoplasms | interventions — Respiratory Rate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telemedicine-Supported Prehabilitation and Rehabilitation (Experimental): Preoperative Phase:
  Wearable Technology: Smartwatch monitoring steps, heart rate, and activity. Physical Exam & Physiotherapy Session: Musculoskeletal evaluation, pelvic floor training via sonographic feedback, posture/respiratory exercises (2-4 weeks pre-surgery).
  Activity Guidelines: Specific daily step targets and exercises to optimize surgical readiness.
  Educational Support: Videos demonstrating pelvic floor training, posture, breathing, and exercises.
  Remote Monitoring & Notifications: Continuous monitoring with inactivity alerts/reminders.
  Online Consultations: Virtual physiotherapy sessions for feedback and plan adjustments.
  Postoperative Phase:
  Physiotherapy Visits: At 3, 4, 6 weeks; 3, 6 months post-surgery for assessment and rehab adjustments.
  Telemonitoring: Continued wearable monitoring, video consultations, and access to educational videos.
  Data Collection: Objective wearable data collected to track progress, adherence, and personalize rehab.
  Interventions: Other: Telemedicine-based prehabilitation and postoperative rehabilitation protocol, including physical activity monitoring, respiratory and postural training, and guidance via telehealth tools.
- Control Group (Standard Preoperative and Postoperative Care) (No Intervention): Preoperative Phase:
  Wearable Technology: Participants receive wearable devices (smartwatch, tablet or phone) for real-time monitoring of physical activity parameters (step count, heart rate, general activity).
  Physical Exam & Physiotherapy: Physiotherapist evaluates musculoskeletal function, provides verbal education on pelvic floor muscle activity, posture, and respiratory exercises; scheduled 2-4 weeks pre-surgery.
  Printed Educational Material: Participants receive printed booklets containing general information, exercises, and activity guidelines to prepare for surgery.
  Telemonitoring (No Notifications): Activity digitally monitored, without sending reminders or prompts for exercise adherence.
  Postoperative Phase:
  Physiotherapy Visits: Scheduled at 3 weeks, 4 weeks, 6 weeks, 3 months, and 6 months post-surgery for progress assessment and rehabilitation adjustments.
  Data Collection: Continuous collection of objective data from wearable devices compared to intervention group.

INTERVENTIONS:
Other: Telemedicine-based prehabilitation and postoperative rehabilitation protocol, including physical activity monitoring, respiratory and postural training, and guidance via telehealth tools. — A combination of wearable technology, activity guidelines, educational support, remote monitoring with notifications and consultations with physiotherapists.
  Arms: Telemedicine-Supported Prehabilitation and Rehabilitation

SUMMARY:
The study titled " The effectiveness of telemedicine monitoring prehabilitation in prostate cancer patients undergoing radical prostatectomy " investigates the impact of a structured telemedicine-supported prehabilitation and rehabilitation program on reducing postoperative urinary incontinence in patients with localized prostate cancer. Radical prostatectomy, a common treatment for localized prostate cancer, is often associated with complications such as urinary incontinence, which significantly affects quality of life. This study aims to address this issue by enhancing patients' physical conditioning and adherence to pre- and postoperative rehabilitation through the use of wearable devices and remote physiotherapy consultations.

DETAILED DESCRIPTION:
Participants in the intervention group will receive a comprehensive prehabilitation program starting 30 -14 days before surgery. They will be equipped with wearable devices (smartwatch and tablet/mobile phone) to monitor physical activity, including parameters like step count and heart rate, allowing for tailored exercise regimens focused on specific daily activity goals. These participants will also have access to educational videos and online consultations with physiotherapists for ongoing support. The program is designed to optimize physical readiness for surgery and improve postoperative recovery outcomes, with continuous monitoring and notifications provided to encourage adherence to the prescribed activities. The control group will receive printed educational materials with general preoperative exercise guidance. This group will have digital monitoring of physical activity, but patients will not receive any reminders or prompts to complete their exercises, they will not have access to online consultations. The primary endpoint of the study is the reduction of urinary incontinence as measured by the 24-hour pad test at 30 days before the surgery and 6 weeks, 3 and 6 months post-surgery. Secondary endpoints include assessments of physical fitness, quality of life, respiratory and postural function, and adherence to the rehabilitation protocol. Both groups will follow structured postoperative follow-ups with physiotherapists at defined intervals to monitor recovery progress and adjust the rehabilitation protocol as necessary. The study spans approximately 6 months for each participant, aiming to generate critical insights into the benefits of telemedicine in enhancing surgical recovery and improving patient outcomes in prostate cancer treatment.

ELIGIBILITY:
Inclusion criteria:

* Biopsy-confirmed localized prostate cancer (ICD code C.61).
* Indicated for radical prostatectomy, with or without pelvic lymphadenectomy (ePLND).
* Not previously treated for prostate cancer, including radiation therapy to the pelvis, major pelvic surgery, or placement of a penile implant or artificial urinary sphincter.
* No known urethral stricture or colostomy or chronic urinary catheterization.
* No medical or current psychiatric disorders that precludes their participation in the study.
* Status of the musculoskeletal system allowing physical exercise.
* Urinary continent at baseline.
* Has reliable internet and the skills/knowledge to use technologies use for the study.

Exclusion criteria:

* Other malignant tumors, except for benign skin carcinoma.
* Active treatment for other oncological diagnoses.
* Presence of preoperative urinary incontinence.
* Diagnosed mental or cognitive disorders.
* Prior pelvic radiotherapy or hormone therapy for prostate cancer recurrence.
* Severe musculoskeletal disorders preventing active exercise
* Inability to use required technologies

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Early Postoperative Incontinence | Baseline evaluated at 30 days before surgery. Evaluated at 6 weeks, 3 months, and 6 months post-surgery.
  Measured by the 24-hour pad weight test.
Time to full Continence Recovery | 3 - 6 months post-surgery
  Time to achieve full continence following surgery (no pads)
Six-Minute Walk Test Distance | 2 weeks pre-surgery, 3 months and 6 months post-surgery
  Distance that a participant is able to walk in 6 minutes on a hard, flat surface.
  Unit of Measure: Meters
Balance Test Composite Score | 2 weeks pre-surgery, 3 months and 6 months post-surgery
  Score from a standardized balance assessment (Berg Balance Scale). Higher scores indicate better balance.
  Unit of Measure: Score Range: 0-56
Lower Limb and abdominal Muscle Strength (Isometric) | 2 weeks pre-surgery, 3 months and 6 months post-surgery
  Isometric strength of targeted muscle groups measured using dynamometer.
  Unit of Measure: Newtons (N)

SECONDARY OUTCOMES:
EPIC-CP Total Score | Baseline (30 days before surgery), 6 weeks, 3 months, and 6 months post-surgery
  Patient-reported outcome measuring health-related QoL in domains relevant to prostate cancer, using the EPIC-CP (Expanded Prostate Cancer Index Composite for Clinical Practice) questionnaire. Higher scores indicate worse QoL.
  Unit of Measure: Score (0-60)
EQ-5D-5L Index Score | Baseline (30 days before surgery), 6 weeks, 3 months, and 6 months post-surgery
  EuroQol (Quality of Life)-5 Dimensions
  Health status measure based on five dimensions of functioning. Score derived using country-specific value sets. Higher scores represent better health status.
  Unit of Measure: Score (range: -0.59 to 1)
Forced Expiratory Volume in One Second (FEV1) | 2 weeks pre-surgery, 3 and 6 months pos-surgery
  FEV1 represents the volume of air that can be forcibly exhaled in the first second of a forced breath. Measurements will be performed using calibrated spirometry according to ERS guidelines. FEV1 is a standard measure of pulmonary function. Higher values indicate better lung function.
  Unit of Measure: Liters
Maximal Voluntary Ventilation (MVV) | 2 weeks pre-surgery, 3 months post-surgery, and 6 months post-surgery
  MVV is the maximum amount of air a participant can inhale and exhale within a specific time frame (12 seconds), extrapolated to one minute. Testing will be conducted using standard spirometry under ERS guidelines. MVV reflects respiratory muscle endurance and ventilatory capacity.
  Unit of Measure: Liters/minute
Daily Step Count | 2 weeks pre-surgery, 3 months and 6 months post-surgery
  Average number of steps recorded per day using a wearable device.
  Unit of Measure: Steps/day
Daily Physical Activity Duration | 2 weeks pre-surgery, 3 and 6 months post-surgery
  Average duration of physical activity (e.g., moderate to vigorous activity) recorded per day using wearable device.
  Unit of Measure: Minutes/day

CONTACTS AND LOCATIONS:
Locations (1):
- Urology clinic, University hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Undecided